CLINICAL TRIAL: NCT03124615
Title: Effect of Enzalutamide Dose Reduction on Fatigue, Cognition, and Drug Trough Levels in Patients With Prostate Cancer
Acronym: EFFECT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGMQ201502
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: Patients will have commenced standard dose enzalutamide (160mg) daily and dose will be reduced if Grade 3 fatigue or cognition change has occurred and if toxicity is attributed to enzalutamide
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enzalutamide (Experimental): Patients will have commenced standard dose enzalutamide (160mg) daily and dose will be reduced if Grade 3 fatigue or cognition change has occurred and if toxicity is attributed to enzalutamide
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide is a FDA and Therapeutic Goods Administration (TGA, Regulatory Authority of therapeutic goods in Australia) approved treatment for castration resistant prostate cancer
  Other Names: Xtandi

SUMMARY:
The primary purpose of this trial is to determine whether dose reduction of enzalutamide in patients with grade 3 fatigue and/or cognition change will lead to an improvement in symptoms while maintaining active drug levels.

Patients within 3 months of starting enzalutamide will be assessed by their oncologist as being potentially eligible for dose reduction due to the onset of moderate to severe fatigue and/or cognition change, which is assessed as being due to enzalutamide

ELIGIBILITY:
Inclusion Criteria:

1. Patients with prostate cancer who have commenced enzalutamide within 3 months
2. Patient must have concomitant LHRH agonist or antagonist (no single agent enzalutamide)
3. Receiving enzalutamide before or after docetaxel
4. Patients may have hormone-sensitive or castrate resistant disease
5. Patients may have metastatic (M1) or non-metastatic (M0) disease
6. Onset of grade 3 or more cognition change and/or fatigue after commencement of enzalutamide considered to be due to enzalutamide

Exclusion Criteria:

1. Clinical dementia
2. Concomitant use of drugs known to impair cognition such as benzodiazepines or antihistamines.
3. Concomitant use of strong CYP3A4 and/ or CYP2C8 inducers or inhibitors.
4. Patient expected to have a change in opioid dose during the study period or have had a change 4 weeks before study entry.
5. Diagnosed with sleep apnoea
6. Brain metastases, prior seizures, drugs that significantly reduce seizure threshold.
7. Active infection or other intercurrent illness that may contribute to fatigue or cognition change within 4 weeks of study entry.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The trial involves only the male population with prostate cancer
Enrollment: 47 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who have an improvement in cognition/ fatigue symptoms | 1 year post enrolment
  The primary endpoint is an improvement in the fatigue and cognition symptoms. Improvement will be de ned as the patient answering 'Better' in the cognition/ fatigue question at the lowest dose of enzalutamide.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Gurney, Principal Investigator — Medical Oncologist
Locations (1):
- Macquarie University, North Ryde, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No